CLINICAL TRIAL: NCT03605563
Title: Changes in the Muscle Tone of Affected Muscle After Fu's Subcutaneous Needling on the Myofascial Trigger Points - a Sample of Lateral Epicondylitis
Brief Title: Fu's Subcutaneous Needling on the Myofascial Trigger Points: Lateral Epicondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Wei Chou, Minister of Rehabilitation, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH107-REC2-019
Record Dates: First submitted 2018-07-18; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Lateral Epicondylitis
Keywords: Fu's subcutaneous needling (FSN); Myofascial trigger point
MeSH Terms: conditions — Tennis Elbow | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FSN: Fu's subcutaneous needling (Experimental): In this arm, the subjects will receive the intervention of FSN on Day1, Day2 and Day4, in total 3 treatments and will be arrange to take efficacy two assessment on Day8 and Day15, separately.
  Interventions: Procedure: Fu's subcutaneous needling
- TENS: Transcutaneous Electric Nerve Stimulation (Active Comparator): In this arm, the subjects will receive the intervention of TENS on Day1, Day2 and Day4, in total 3 treatments and will be arrange to take efficacy two assessment on Day8 and Day15, separately.
  Interventions: Procedure: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Procedure: Fu's subcutaneous needling — Fu's Subcutaneous Needle (FSN), is an innovation for the treatment of myofascial pain and trigger points. The needle is a non-injection needle, and the fact that both needles are manipulated and act on soft connective tissue.
  FSN abstains from the muscle and deep fascia layers and is confined to only the subcutaneous layer where collagen fibers are most abundant. As the subcutaneous layer is poorly innervated, pain is less than other needling therapies.
  FSN is also currently being used successfully to treat non-musculoskeletal conditions.
  Arms: FSN: Fu's subcutaneous needling
Procedure: Transcutaneous electrical nerve stimulation — Transcutaneous electrical nerve stimulation (TENS or TNS) is the use of electric current produced by a device to stimulate the nerves for therapeutic purposes.
  TENS, by definition, covers the complete range of transcutaneously applied currents used for nerve excitation although the term is often used with a more restrictive intent, namely to describe the kind of pulses produced by portable stimulators used to treat pain. The unit is usually connected to the skin using two or more electrodes. A typical batteryoperated TENS unit is able to modulate pulse width, frequency and intensity. Generally TENS is applied at high frequency (>50 Hz) with an intensity below motor contraction (sensory intensity) or low frequency (<10 Hz) with an intensity that produces motor contraction.
  Arms: TENS: Transcutaneous Electric Nerve Stimulation

SUMMARY:
Lateral epicondylitis, also called tennis elbow, is the most common disease in elbow-pain symptoms. The symptoms can have a major impact on the patient's activity of daily life, including turning a doorknob, lifting a full coffee cup to mouth, or wringing out a dish rag.

This is a randomized study, the investigators will evaluate the immediate, short-term, and long-term effect of Fu's subcutaneous needling on the patients suffering with lateral epicondylitis.

DETAILED DESCRIPTION:
Lateral epicondylitis, also called tennis elbow, is the most common disease in elbow-pain symptoms. The major mechanism is overuse of the flexors, extensors and supination muscles in the wrist, causing micro-trauma in the muscles attachment to the lateral epicondyle of the elbow. The long-term accumulated and poor repaired trauma causes myofascial trigger points in the related muscles. Patients often describe pain at the lateral aspect of the elbow. Pain can be further elicited with passive wrist flexion and by resisting active wrist extension. Symptoms also include weakness in the grip strength and limitation of elbow motion. Therefore, it can have a major impact on the patient's activity of daily life, including turning a doorknob, lifting a full coffee cup to mouth, or wringing out a dish rag.

Fu's subcutaneous needling (FSN), as one of the dry needle treatments, performed by swaying a disposable Fu's subcutaneous needle parallel to the underlying muscles after penetrating the skin to the subcutaneous fascia. With the reperfusion activities, myofascial pain and soft tissue pain caused by myofascial trigger points can be decreased effective simultaneously. So far, there is no solid research or clinical trial to evaluate the efficacy of the treatment yet.

The investigators will conduct the randomized experiment to evaluate the immediate, short-term, and long-term effect of FSN. The outcome measures include visual analog scale, patient-rated tennis elbow evaluation questionnaire, pressure pain threshold, pain-free grip test, muscle tone changes and ultrasonographic evaluaton of the common extensor tendon.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects older than 20 years of age who can cooperate with the experimental volunteers.

  2. Suffering from epicondylitis of the humerus for more than one month, and subjective pain intensity (VAS) greater than 5 points.

  3. There is a local tender point at the upper elbow of the elbow, and the isometric resistance test of the forearm to make a spin will induce pain.

  4. Under soft tissue ultrasound, the thickness of the common tendon of the extensor carpi muscles is more than 0.15 mm greater than that of the healthy side.

Exclusion Criteria:

* 1. There are contraindications to general treatment, such as serious medical problems, recent serious trauma, or pregnant women.

  2. There has been a history of drug abuse (including excess alcohol) that affects pain assessors.

  3. Have received neck, upper back, or upper and lower limb surgery. 4. People with central or peripheral nerve disease. 5. Cognitive impairment, unable to cooperate with the experimenter. 6. Patients currently receiving other treatments for epicondylitis of the humerus.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-04-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scales | 1 day
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.

SECONDARY OUTCOMES:
Pressure Pain Threshold | 1 day
  Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain. This measure has proven to be commonly useful in evaluating tenderness symptom.
Myotone of MTrPs | 1 day
  Muscle tone is the muscle's resistance to passive stretch during resting state. Myotone will help the investigators to get muscle parameters such as tone, elasticity and stiffness.
Pain-free grip test | 1day
  The pain-free grip (PFG) test is used to measure the amount of force that the patient generates to the onset of pain; when there is no pain the test result could be regarded as maximum grip strength. It is commonly performed in patients with lateral epicondylalgia (LE). LE is characterised by the presence of pain over the lateral humeral epicondyle which is provoked by at least two of: gripping, resisted wrist or middle finger extension, or palpation (Stratford et al 1993) in conjunction with reduced PFG over the affected side (Stratford et al 1993; Vicenzino et al 1996; Vicenzino et al 1998).

CONTACTS AND LOCATIONS:
Overall Officials: Li-Wei Chou, PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang CH, Lin CY, Sun MF, Fu Z, Chou LW. Efficacy of Fu's Subcutaneous Needling on Myofascial Trigger Points for Lateral Epicondylalgia: A Randomized Control Trial. Evid Based Complement Alternat Med. 2022 Mar 14;2022:5951327. doi: 10.1155/2022/5951327. eCollection 2022. PMID 35321501